CLINICAL TRIAL: NCT06803953
Title: Definition of a Cut Off Value for S.P.A.T (Skin Prick Automated Test) Device Corresponding With Sensitisation to Both Birch and House Dust Mite Allergens, in Allergic Subjects
Brief Title: Evaluation of an Adjusted Cutoff Value for S.P.A.T (Skin Prick Automated Test) Device in Allergic Subjects
Acronym: SPATprovocatio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hippocreates (Industry)
Collaborators: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HIP-001
Record Dates: First submitted 2025-01-03; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: House Dust Mite Allergy; Birch Pollen Allergy
MeSH Terms: conditions — Dust Mite Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HDM allergic patients (Experimental): HDM allergic patients receive a nasal allergen provocation test with house dust mite allergens (der p and der f) to confirm the clinical relevance of the allergy.
  All patients receive a conventional skin prick test on the one arm and an automated test on the other arm.
  Interventions: Device: Skin Prick Automated Test; Diagnostic Test: Skin Prick Manual Test; Diagnostic Test: Nasal Allergen Challenge
- Birch pollen allergic patients (Experimental): Birch pollen allergic patients receive a nasal allergen provocation test with birch allergen (bet v) to confirm the clinical relevance of the allergy.
  All patients receive a conventional skin prick test on the one arm and an automated test on the other arm.
  Interventions: Device: Skin Prick Automated Test; Diagnostic Test: Skin Prick Manual Test; Diagnostic Test: Nasal Allergen Challenge
- Non allergic patients (Experimental): Non allergic patients did not receive a nasal allergen provocation test. All patients receive a conventional skin prick test on the one arm and an automated test on the other arm.
  Interventions: Device: Skin Prick Automated Test; Diagnostic Test: Skin Prick Manual Test

INTERVENTIONS:
Device: Skin Prick Automated Test — skin prick test to detection sensitisation to aeroallergens
Diagnostic Test: Skin Prick Manual Test — skin prick test to detection sensitisation to aeroallergens
Diagnostic Test: Nasal Allergen Challenge — nasal allergen challenge with either house dust mite allergens or birch pollen allergens
  Arms: Birch pollen allergic patients; HDM allergic patients

SUMMARY:
Skin prick test (SPT) is a first line diagnostic test to detect type I hypersensitivity in patients suspected of an inhalant allergy. A novel S.P.A.T. or Skin Prick Automated Test device has been developed to enable more standardised allergy testing. In two independent studies, Gorris and colleagues previously showed that test results after S.P.A.T. are less variable and more consistent compared to conventional skin prick testing (Gorris et al. Allergy. 2023; Seys et al. Rhinology 2024). In these studies conducted in volunteers, a cutoff value of 4.5 mm has been proposed based on the 97.5 percentile level of glycerol control wheals.

The current study aims to determine a cutoff value corresponding to the highest accuracy to discriminate between sensitized-allergic and non sensitized, non allergic subjects for both house dust mite and birch allergens.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent signed by study patient and investigator;
* Subjects with Health Social Identification Number;
* Allergic subjects with rhinitis with or without asthma and with or without conjunctivitis symptoms with proof of sensitisation to an inhalant allergy, either house dust mite ( Dermatophagoides pteronyssinus) or birch pollen by a positive skin prick test (SPT) with a wheal diameter ≥3 mm as compared to negative control. The clinical response against the culprit allergen will be assessed by a positive nasal allergen provocation test. (patients must not have clinical symptoms corresponding to both sensitization).
* Non-allergic subjects with proof of lack of sensitisation to any of the above referred allergens by a negative conventional skin prick test less than 2 years.
* Normal lung function as judged by investigator with FEV 1 and FEV 1/FVC ≥ 70% of predicted
* Willing and able to comply with clinic visits and study-related procedures;
* Able to understand and complete study-related questionnaires.

Exclusion Criteria:

* Skin pathology like chronic or exuberant urticaria, dermographism, chronic dermatitis that needs daily treatment;
* Any skin abnormalities, which could negatively - in the opinion of the investigator - affect the test results, including large scars and tattoos on the forearm ;
* Patients with clinical symptoms corresponding to both sensitization to birch and house dust mite
* Use of antihistaminic medication < 7 days before the start of the study;
* Use of tricyclic antidepressants (antihistamine activity) < 7 days before the start of the study;
* Use of topical (on the forearm) or systemic corticoids < 7 days before the start of the study;
* Use of any monoclonal antibodies such as omalizumab, dupilumab, mepolizumab < 6 months before the start of the study;
* Use of oral systemic corticosteroids within 4 weeks prior to screening
* Use of intramuscular systemic corticosteroids within 3 months prior to screening
* Use of allergen immunotherapy for the allergen tested (<2 y) or another inhalant allergen;
* Pregnancy or breastfeeding;
* Women without highly effective contraception (hormonal contraception, intrauterine device, bilateral tubal occlusion/ligation, vasectomized partner, sexual abstinence) at least one month prior to inclusion and during the study;
* Incapacitated subjects;
* Subjects who do not speak the local language (French);
* Subjects who cannot read or write.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Cutoff value with highest accuracy based on longest wheal diameter after SPAT | 15 minutes after SPAT
  The cutoff value that corresponds to the highest F1 score of the accuracy of S.P.A.T. to detect sensitisation to both house dust mite and birch allergens by measuring the longest diameter of wheal size.

SECONDARY OUTCOMES:
Accuracy of SPAT compared to conventional SPT | 15 minutes after SPAT
  The non-inferiority of the accuracy of S.P.A.T. compared to the conventional SPT to detect sensitisation for both house dust mite and birch allergens in allergic and non-allergic subjects will be evaluated by comparing the F1 score of SPT and SPAT, measuring the longest diameter of wheal size.

OTHER OUTCOMES:
Intensity of allergy symptoms | 15 minutes after SPAT
  The intensity of allergy symptoms will be evaluated by Lebel score and compared to wheal size after positive SPT.
Intensity of allergy symptoms | 15 minutes after SPAT
  The intensity of allergy symptoms will be evaluated by PNIF measurement and compared to wheal size after positive SPT.
Longest wheal diameter measurement through S.P.A.T. web viewer compared to conventional ruler-based measurement | 15 minutes after SPAT
  The concordance of wheals' size measurement by the S.P.A.T. web viewer and investigator/ trained and qualified staff member will be evaluated by correlation analysis.
Time to perform skin prick test | at time of SPAT
  The time to perform SPAT and conventional SPT will be evaluated by timing the duration between the start of executing the test and the end of the reading of the test (without timing the 15 minutes of waiting before reading).
Longest wheal diameter with S.P.A.T. compared to average diameter with conventional SPT | 15 minutes after SPAT
  The longest diameter of wheal size measured with S.P.A.T. will be compared to the average (D+d/2) and the longest diameter of wheal size measured by conventional SPT.
Cutoff value with highest accuracy based on wheal area | 15 minutes after SPAT
  For the S.P.A.T., a cutoff value will be calculated similar to above by using the wheal area evaluated by F1 score.
Accuracy of SPAT based on wheal area compared to conventional SPT | 15 minutes after SPAT
  The non-inferiority of S.P.A.T accuracy using the wheal area compared to conventional SPT longest wheal diameter will be evaluated comparing the F1 score.
Cutoff with highest accuracy based on histamine equivalent prick index | 15 minutes after SPAT
  For the S.P.A.T., the HEP (histamine equivalent prick) index based on the wheal diameter and wheal area will be calculated. The cut-off value will be calculated similar to above. The HEP index is defined as allergen induced area/ histamine induced area or allergen induced diameter/histamine induced diameter.
Accuracy of SPAT based on histamine equivalent prick index compared to conventional SPT | 15 minutes after SPAT
  The non-inferiority of accuracy using the HEP-index compared to conventional SPT longest wheal diameter will be evaluated comparing the F1 score.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Gherasim, MD, Principal Investigator — Alyatec
Locations (1):
- Alyatec, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided